CLINICAL TRIAL: NCT04171154
Title: The Effects of Brief, Psychological Interventions (Micro-Interventions) on the Individual Stress Reactivity
Brief Title: Effects of Micro-Interventions on Stress Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-54k
Record Dates: First submitted 2019-11-08; First posted 2019-11-20 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Psychological Stress; Physiological Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expectation (Experimental): Participants are asked to think of three strength which have helped them in prior stressful events. They then have to think of ways how these strength may help them in future stressful situations, i.e. a test in this experiment.
  Interventions: Behavioral: Expectation
- Acceptance (Experimental): Participants listen to an audio-instruction on cognitive defusion. They shall observe the thoughts and feelings of stress and, with the help of the instruction, distance themselves from it.
  Interventions: Behavioral: Acceptance
- Control (No Intervention): Participants wait for the stress-test to start.

INTERVENTIONS:
Behavioral: Expectation — writing task
  Arms: Expectation
Behavioral: Acceptance — listening
  Arms: Acceptance

SUMMARY:
This study aims to investigate the effects of short, psychological interventions on bio-psychological stress responses after an acute stressor. The efficacy of two different approaches (expectation-bases vs. acceptance-based) will be compared to a control-group.

ELIGIBILITY:
Inclusion Criteria:

* fluent in German language

Exclusion Criteria:

* chronic disease
* mental disease
* the evening before the day of the experiment until end of the experiment (the next day):
* caffeine, alcohol, intensive physical exercise, chewing gum
* acute hay fever
* current intake of psychotropic medication
* current intake of orale contraceptives
* visual impairments
* heart conditions (self and close relatives)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Change in Subjective Stress Ratings | at baseline, before the intervention, after the intervention; during the stressor, after the stressor; in total 45 minutes
  VAS (visual analogue scale)
Change in Cortisol Levels | at baseline (min. -37), after the intervention (min. -19), after the stressor (min. 0), recovery 1 (min. +15), recovery 2 (min. +30); in total 67 minutes
  saliva sample
Changes in Heart-Rate-Variability (HRV) | during baseline (duration 10 minutes), during the stressor (duration 20 minutes), during recovery (duration 10 minutes); in total 40 minutes
  electrocardiogram
Changes in Affect | at baseline, after the stressor; in total 45 minutes
  VAS (visual analogue scale)

SECONDARY OUTCOMES:
Self-Efficacy | at baseline, after the recovery-phase; in total 55 minutes
  questionnaire (self-efficacy scale; Schwarzer & Jerusalem, 1999)
Positivity | at baseline, after the recovery-phase; in total 55 minutes
  questionnaire (positivity scale; Caprara et al., 2012, König, 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Euteneuer, Prof. Dr., Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps University Marburg Medical Center, Marburg, Germany